CLINICAL TRIAL: NCT07264582
Title: A Citizen Science Approach to Increase HIV/STI/HCV Testing and Substance Use Service Utilization Among Survivors of Sex Trafficking Living in New York City
Brief Title: HIV/STI/HCV Testing and Overdose Prevention Among Survivors of Sex Trafficking
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Alissa Davis, Associate Professor, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: AAAV8351; 1R34DA063049 (NIH)
Record Dates: First submitted 2025-11-19; First posted 2025-12-04 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: HIV Testing; STI; HCV; Overdose, Drug
Keywords: HIV; STI; HCV; overdose prevention; crowdsourcing; citizen science
MeSH Terms: conditions — Sexually Transmitted Diseases; Drug Overdose

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive the digital crowdsourced messaging materials or existing HIV/STI/HCV testing and overdose prevention materials. The investigators will examine the effects of the intervention on increasing HIV/STI/HCV testing and increasing utilization of overdose prevention kits.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Crowdsourced Messaging Intervention (Experimental): The digital crowdsourced intervention will be presented to participants in the intervention arm.
  Interventions: Behavioral: Sex Trafficking Survivor-Developed Digital Crowdsourced Intervention
- Standard of Care (No Intervention): Standard informational materials about HIV/STI/HCV testing and overdose prevention currently used by Departments of Health and other health organizations will be presented to participants in the control arm.

INTERVENTIONS:
Behavioral: Sex Trafficking Survivor-Developed Digital Crowdsourced Intervention — Survivors of sex trafficking will participate in crowdsourcing contests to create digital materials to promote HIV/STI/HCV testing and use of overdose prevention kits. Entries will be judged by community and expert judges. Top entries will be selected for the digital intervention and presented to participants in the intervention arm.
  Arms: Crowdsourced Messaging Intervention

SUMMARY:
This project will assess whether a digital survivor crowdsourced intervention can increase HIV/STI/HCV testing and overdose prevention kit utilization among survivors of sex trafficking living in New York City. Survivors of sex trafficking have among the highest rates of HIV/STIs/HCV and substance use disorder (SUD), yet they face substantial barriers to care, including lack of information about care and financial and logistical constraints. In addition, there is a lack of public health messaging tailored specifically for survivors of sex trafficking to meet their needs. Citizen science approaches, such as crowdsourcing (i.e., engaging groups of individuals to address public health challenges and share solutions), are scalable, cost-effective tools that can increase HIV/SUD prevention and treatment utilization. Crowdsourcing can be used to engage survivors in developing tailored messaging to promote HIV/STI/HCV testing, overdose prevention, and treatment utilization. Complementing crowdsourcing, specimen self-collection with remote HIV/STI/HCV testing and online delivery of overdose prevention kits to survivors may also increase use of needed healthcare services. Study aims are: 1) develop crowdsourced digital messages to promote HIV/STI/HCV testing uptake and utilization of overdose prevention services for substance use among sex trafficking survivors; 2) in a randomized controlled trial, to compare the survivor-crowdsourced HIV and substance use intervention to existing public health messaging among sex trafficking survivors (n=368) in New York City; and 3) assess the contribution of multi-level factors on reach, effectiveness, adoption, implementation, and maintenance (RE-AIM) outcomes. This work will result in a digital crowdsourced intervention to increase HIV/STI/HCV testing uptake, overdose prevention kit utilization, and linkage to care among survivors of sex trafficking. This project will also result in a crowdsourcing and messaging toolkit that can be broadly distributed to public health and other agencies across the country for their use in designing messaging campaigns for survivors. Findings from this project will lay the groundwork for citizen science-developed HIV and SUD interventions for sex trafficking survivors across the US.

DETAILED DESCRIPTION:
The investigators propose to develop and assess whether a digital survivor-crowdsourced (i.e., engaging individuals to address public health challenges and share solutions) intervention can increase testing for HIV, sexually transmitted infections (STIs), and hepatitis C virus (HCV) and the utilization of life-saving overdose prevention practices and services among survivors of sex trafficking (ST) in New York City (NYC). ST survivors have higher risk substance use (e.g., injection drug use, fentanyl) than women who are not trafficked -- >84% have used substances, with ~33% experiencing forced substance use, and ~70% a drug overdose. ST survivors have higher HIV/STI prevalence rates (up to 70%) than even non-trafficked women in sex work. Nearly 50% of survivors have branding tattoos, increasing their risk for HCV. Despite their elevated rates of HIV/STIs/HCV and substance use disorder (SUD), there is a lack of public health messaging tailored specifically for ST survivors, and much of the existing messaging is denigrating toward this population. Survivors also face substantial barriers to care, including lack of information about care access and logistical constraints. In the absence of innovative interventions tailored for this population, health problems among ST survivors will persist.

The Study's Specific Aims are:

Aim 1: Develop crowdsourced digital messages to promote HIV/STI/HCV testing uptake and utilization of overdose prevention services for substance use among female ST survivors. To achieve this aim, in partnership with our Citizen Collaborative Research Board (CCRB), the investigators will use in-depth interviews and conduct a series of designathons, launched via a national crowdsourcing open call, in which survivors ideate, prototype and present multimedia content to promote HIV/STI/HCV testing uptake and utilization of overdose prevention services among peers.

Aim 2: In a randomized controlled trial, to compare the survivor-crowdsourced HIV and substance use intervention to existing public health messaging among ST survivors (n=368) in New York City.

Hypothesis: The crowdsourced intervention will increase HIV/STI/HCV testing uptake and utilization of overdose prevention services among survivors compared to control content. The primary outcome will be online HIV/STI/HCV tests completed and online ordering of overdose prevention kits. Secondary outcomes will be linkage to HIV/STI/HCV care, PrEP, and substance use disorder (SUD) services.

Aim 3: Assess the contribution of multi-level factors on reach, effectiveness, adoption, implementation, and maintenance (RE-AIM) outcomes. The investigators will use the PRISM framework and a mixed methods approach to assess RE-AIM outcomes via qualitative interviews, surveys, and HIV/STI/HCV testing and overdose prevention kit referral vouchers.

Hypothesis: HIV/STI/HCV testing and overdose prevention kit referral and uptake will be significantly greater among the crowdsourced intervention arm than among the control arm.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Born biologically female or identify as a woman
* Living in New York City
* Used illicit substances within the past 12 months or has a history of substance use dependency
* Would feel safe participating in the study
* Is a survivor of sex trafficking as defined by the following criteria: 1) Has the individual ever had sex for things of value? If 'Yes', then the individual must also answer 'Yes' to the following question, 2) Was the individual pressured or forced by another person to do this?

Exclusion Criteria:

* Not willing to provide consent or not able to understand study procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
HIV/STI/HCV testing uptake | From baseline to the 6 month follow-up
  The number of participants who ordered and returned a HIV/STI/HCV test kit from baseline to the 6-month follow-up. It is a dichotomous outcome (yes/no).
Overdose Prevention Kit Uptake | From baseline to the 6 month follow-up
  The number of participants who ordered an overdose prevention kit from baseline to the 6-month follow-up. It is a dichotomous outcome (yes/no).

SECONDARY OUTCOMES:
Linkage to HIV/STI/HCV care | From baseline to the 6-month follow-up
  The number of participants who test positive for HIV/STI/HCV and who access care. It is a dichotomous outcome (yes/no).
Linkage to substance use services | From baseline to the 6 month follow-up
  The number of participants who use substances who accessed substance use services from baseline to the 6-month follow-up. It is a dichotomous outcome (yes/no).
HIV/STI stigma | Baseline, 3 months, and 6 months
  Mean score change in stigma from baseline to 3 months follow-up and 6 months follow-up. Higher scores correspond to higher stigma levels.
Substance use stigma | Baseline, 3 months, and 6 months
  Mean score change in stigma from baseline to 3 months follow-up and 6-months follow-up. Higher scores correspond to higher stigma levels.

CONTACTS AND LOCATIONS:
Overall Officials: Alissa Davis, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Survey data from baseline and follow-up assessments will be preserved and deposited in the National Addiction and HIV Data Archive Program (NAHDAP) repository.
Supporting Information: Study Protocol, SAP
Time Frame: Final submission and release of the study data will occur within 12 months following publication of the main outcomes paper and will be available through the National Addiction and HIV Data Archive Program (NAHDAP) repository in perpetuity.
Access Criteria: Data will be deposited as a restricted use dataset in NAHDAP. Investigators interested in analyzing the data must submit a request to NAHDAP and receive approval before they will be able to access the data.